CLINICAL TRIAL: NCT04701645
Title: Pilot Study of an Implantable Microdevice for Evaluating Drug Responses in Situ in Ovarian, Fallopian Tube, and Peritoneal Cancer
Brief Title: Microdevice In Ovarian, Fallopian Tube, And Peritoneal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Oliver Jonas, sponsor, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-357; R21CA216796 (NIH)
Record Dates: First submitted 2020-10-08; First posted 2021-01-08 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Ovarian Cancer Stage III; Ovarian Cancer Stage IV; Fallopian Tube Cancer Stage IV; Fallopian Tube Cancer Stage III
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Implantable Microdevice; Ovarian Cancer Stage III; Ovarian Cancer Stage IV; Fallopian Tube Cancer Stage IV; Fallopian Tube Cancer Stage III
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1: Primary cytoreduction (Experimental): Patients with a new or suspected diagnosis of ovarian cancer who are deemed surgical candidates for primary cytoreductive surgery (as per their surgical gynecologic oncologist) and who have not yet undergone surgery.
  * Participants will undergo percutaneous placement of several microdevices in a selected tumor deposit prior to surgery.
  * The microdevices will dwell in the tumor tissue for approximately 24 +/- 8 hours to allow time for tissue effects of the drugs in the microdevice reservoirs. Microdevices will then be removed by resection of the tumor mass during a previously planned, and clinically indicated, surgical procedure.
  Interventions: Combination Product: Microdevice
- Cohort 2: Surgical assessment for primary surgery (Experimental): Patients with newly diagnosed ovarian cancers who are being considered for either primary surgery or neoadjuvant chemotherapy by their surgical gynecologic oncologist, and who require a laparoscopic procedure to determine their candidacy for surgery.
  * Participants will undergo percutaneous placement of several microdevices in a selected tumor deposit prior to surgery.
  * The microdevices will dwell in the tumor tissue for approximately 24 +/- 8 hours to allow time for tissue effects of the drugs in the microdevice reservoirs. Microdevices will then be removed by resection of the tumor mass during a previously planned, and clinically indicated, surgical procedure.
  Interventions: Combination Product: Microdevice
- Cohort 3: Secondary cytoreduction (Experimental): Patients with recurrent ovarian cancer who are candidates for secondary cytoreduction, e.g.to confirm diagnosis of recurrent ovarian cancer and/or remove oligometastatic lesions.
  * Participants will undergo percutaneous placement of several microdevices in a selected tumor deposit prior to surgery.
  * The microdevices will dwell in the tumor tissue for approximately 24 +/- 8 hours to allow time for tissue effects of the drugs in the microdevice reservoirs. Microdevices will then be removed by resection of the tumor mass during a previously planned, and clinically indicated, surgical procedure.
  Interventions: Combination Product: Microdevice
- Cohort 4: Interval debulking surgery following neoadjuvant chemotherapy (Experimental): Patients with newly diagnosed ovarian cancers who have undergone neoadjuvant chemotherapy and are deemed surgical candidates for interval debulking surgery (as per their surgical gynecologic oncologist) and who have not yet undergone surgery.
  * Participants will undergo percutaneous placement of several microdevices in a selected tumor deposit prior to surgery.
  * The microdevices will dwell in the tumor tissue for approximately 24 +/- 8 hours to allow time for tissue effects of the drugs in the microdevice reservoirs. Microdevices will then be removed by resection of the tumor mass during a previously planned, and clinically indicated, surgical procedure.
  Interventions: Combination Product: Microdevice

INTERVENTIONS:
Combination Product: Microdevice — Placement of 1 to 6 implantable microdevices with multiple miniature drug reservoirs into a tumor mass 24 +/- 8 hours prior to surgery. Drugs will be released over 24 (+/- 8) hours while the microdevice is in the tumor prior to retrieval. The local tissue is retrieved along with the microdevice and no residual drug will remain.
  * Each microdevice will harbor up to 20 drugs and drug combinations relevant to the treatment of ovarian cancer.
  * Each drug or drug combination will be released from a single, separate reservoir. At least two reservoirs will harbor a drug vehicle only.
  * Drugs will include all or a subset of the following: Cisplatin, Carboplatin, Paclitaxel, Doxorubicin or pegylated liposomal doxorubicin (PLD), Cyclophosphamide, Etoposide, Gemcitabine, Ifosfamide, Pemetrexed, Topotecan, Vinorelbine, Olaparib, Niraparib, Rucaparib, Carboplatin + paclitaxel (combination), Carboplatin + doxorubicin (combination),Carboplatin + gemcitabine (combination)

SUMMARY:
This pilot study will assess the feasibility of using an implantable microdevice to measure local intratumor response to chemotherapy and other clinically relevant drugs in ovarian, fallopian tube, and primary peritoneal cancer.

The name of the study intervention involved in this study is:

-implantable microdevice

DETAILED DESCRIPTION:
This research study will assess the feasibility of using an implantable microdevice to measure local intratumor response to chemotherapy and other clinically relevant drugs in ovarian, fallopian tube, and primary peritoneal cancer.

Participants with suspected or confirmed ovarian cancer whose treatment plan includes surgery as a component of standard-of-care treatment will be identified.

-The research study procedures include screening for eligibility and study treatment including evaluations and follow-up.

The name of the study intervention involved in this study is: implantable microdevice

* Participant will undergo percutaneous placement of several microdevices in a selected tumor deposit prior to surgery. The microdevices will dwell in the tumor tissue for approximately 24 +/- 8 hours to allow time for tissue effects of the drugs in the microdevice reservoirs. Microdevices will then be removed by resection of the tumor mass during a previously planned, and clinically indicated, surgical procedure.
* It is expected that about 20 people will take part in this research study.

This research study is a Pilot Study, which is the first time investigators are examining this microdevice. The FDA (the U.S. Food and Drug Administration) has not approved the microdevice as a tool to identify which cancer treatment is best for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have suspected or confirmed clinically advanced stage (III-IV, defined as disease outside of the pelvis) ovarian, fallopian tube, or peritoneal cancer. If a patient has suspected ovarian cancer but final histologic analysis does not show evidence of ovarian cancer, the patient will be removed from the study and replaced.
* Participants must meet one of the following clinical categories:

  * Cohort 1: Patients with a new or suspected diagnosis of ovarian cancer who are deemed surgical candidates for primary cytoreductive surgery (as per their surgical gynecologic oncologist) and who have not yet undergone surgery.
  * Cohort 2: Patients with newly diagnosed ovarian cancers who are being considered for either primary surgery or neoadjuvant chemotherapy by their surgical gynecologic oncologist, and who require a laparoscopic procedure to determine their candidacy for surgery.
  * Cohort 3: Patients with recurrent ovarian cancer who are candidates for secondary cytoreduction, e.g. to confirm diagnosis of recurrent ovarian cancer and/or remove oligometastatic lesions.
  * Cohort 4: Patients with newly diagnosed ovarian cancers who have undergone neoadjuvant chemotherapy and are deemed surgical candidates for interval debulking surgery (as per their surgical gynecologic oncologist) and who have not yet undergone surgery.
* Participants must be 18 years of age or older.
* Patients must be deemed medically stable to undergo both percutaneous procedures and standard-of-care surgical procedures by their treating gynecologic oncologist and medical oncologist.
* Participants will undergo laboratory testing within 14 days* prior to the microdevice placement.

  * Patients must have absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 75,000/mcL
  * PT (INR) < 1.5
  * PTT < 1.5x control
  * Women of childbearing potential must have negative pregnancy test (urine or serum) **Cohort 4 patients should undergo laboratory testing within 7 days prior to the microdevice placement
* Participants must be evaluated by a surgical gynecologic oncologist who will determine the clinically appropriate treatment strategy (primary surgery or neoadjuvant chemotherapy) based on clinical history and extent of disease. The patient's surgical and/or medical gynecologic oncologist must also confirm the patient's medical fitness to undergo an additional biopsy procedure and the indicated surgical procedure. The patient must have a plan to undergo surgery for clinical purposes.
* The following criteria must be met:

  * Participants must have undergone an abdominal/pelvic CT scan that both assesses the extent of disease and identifies an area of tumor amenable to safe microdevice placement. CT scans with both oral and IV contrast media are preferred but not required.

CT scans performed at outside institutions are acceptable providing that the images are considered adequate to assess the stage of the disease and to assess the safety and feasibility of the placement of the microdevices and their retrieval during standard-of care surgery. CT scan must be completed within 4 weeks prior to the microdevice placement.

* Patient has sufficient volume of disease as measured by CT scan to allow implantation of the microdevice.
* Patient has sufficient volume of disease that removal of the lesion where the microdevice is placed will not potentially affect adequate tissue for diagnosis.
* A lesion can be selected where the microdevice is to be implanted that is

  * Amenable to percutaneous placement
  * Amenable to removal at the time of surgery or laparoscopy. If patient is undergoing laparoscopy, the lesion must be able to be removed using a laparoscopic approach in a manner that would not significantly alter the procedure or affect patient safety, per opinion of the surgical oncologist.

    * Patients must have the ability to understand and the willingness to sign a written informed consent document.
    * Patients must be willing to undergo research-related genetic sequencing (somatic and germline) and data management, including the deposition of de-identified genetic sequencing data in NIH central data repositories.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit the safety of a biopsy and/or surgery.
* Pregnant women are excluded from this study because of the possible increased dose of radiation from imaging associated with the microdevice placement and the potential risk to the pregnancy of the biopsy/device placement in an abdominal lesion.
* Uncorrectable bleeding or coagulation disorder known to cause increased risk with surgical or percutaneous biopsy procedures.
* Significant risk factors (including, but not limited to, high risk of venous thrombosis, pulmonary embolism, stroke or myocardial infarction) precluding the safe cessation of anticoagulation medication as per SIR guidelines. (Patients taking low-dose aspirin only do not need to be excluded.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as defined in the CTCAE v5.0 | Up to 2 months
  Descriptive statistics will be used to evaluate the safety of microdevice placement and removal, including reporting the maximum grade AE by type and organ class with 95% binomial confidence intervals.
Number of implanted microdevices successfully retrieved | Up to 32 hours
  Defined as the ability to retrieve the microdevice with sufficient tissue, of sufficient quality, for downstream histopathology analysis and interpretation of at least 50% of the microdevice reservoirs. For purposes of this endpoint, feasibility will be assessed on a per-device basis rather than a per-patient basis, with each microdevice considered to be relatively independent in terms of placement, retrieval, and analysis.

OTHER OUTCOMES:
Measure local intratumor response to different agents | Up to 32 hours
  Response assessed via apoptotic index measured by immunohistochemistry.
  Inferences will use two-sided alpha = 0.05 and report 95% confidence intervals with any point estimates.
Correlate extent of tumor response with platinum response category | Up to 3 years
  Platinum response category is defined as follows for both initial and secondary platinum exposure: platinum refractory (progression within 2 months of platinum-based chemotherapy), platinum resistant (progression within 2-6 months of platinum-based chemotherapy), and platinum sensitive (progression within 6-12 months of platinum based chemotherapy).
  For dichotomous/categorical tumor features and patient outcomes, we will use Fisher's exact test. For continuous variables we will use a two-sided t-test if the data is approximately normally distributed, and Wilcoxon rank sum test if otherwise.
Correlate extent of tumor response with platinum-free interval | Up to 3 years
  Platinum-free interval is defined as the interval between the date of the last platinum dose and the date of relapse detection.
  For dichotomous/categorical tumor features and patient outcomes, we will use Fisher's exact test. For continuous variables we will use a two-sided t-test if the data is approximately normally distributed, and Wilcoxon rank sum test if otherwise.
Correlate extent of tumor response with progression-free survival | Up to 3 years
  Progression defined using RECIST 1.1 criteria; progression-free survival measured in months.
  For dichotomous/categorical tumor features and patient outcomes, we will use Fisher's exact test. For continuous variables we will use a two-sided t-test if the data is approximately normally distributed, and Wilcoxon rank sum test if otherwise.
Correlate extent of tumor response with exploratory biomarkers of drug response | Up to 32 hours
  Candidate biomarkers for chemotherapy and PARP inhibitor response in ovarian cancer include RAD51 focus formation, markers of DNA damage (e.g. gamma-H2AX), and immune infiltrates. Each biomarker will be evaluated by immunohistochemistry to generate a quantitative score for the number of marker-positive cells per number of cells analyzed. Descriptive statistics will be used to summarize the results for each biomarker across multiple microdevices and drugs.
Compare extent of tumor response to drug among multiple microdevices implanted within a single tumor | Up to 32 hours
  Response will be assessed via apoptotic index measured by immunohistochemistry and will be compared among multiple microdevices implanted within a single tumor.
Correlate extent of tumor response with genetic features of the tumor tissue | Up to 32 hours
  Genetic alterations will be catalogued in terms of single nucleotide variants, insertions/deletions, and copy number changes in individual genes in the tumor tissue. Each alteration will be scored as "present" or "absent" in a tumor. Descriptive statistics will be used to summarize the frequency of each genomic event across multiple microdevices and drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stover, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu